CLINICAL TRIAL: NCT05755646
Title: Feasibility of an RCT to Investigate the Efficacy of Ice Plant Intensive Cream for the Prevention of Hand-foot Syndrome in Patients With Breast Cancer Receiving Therapy With Doxorubicin and/or Docetaxel: Pilot Randomized Controlled Trial
Brief Title: Ice Plant Intensive Cream for the Prevention of Hand-Foot Syndrome in Breast Cancer: Pilot Randomized Controlled Trial
Acronym: WIn-HFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: S00748-NIM
Record Dates: First submitted 2023-01-30; First posted 2023-03-06 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2023-01

CONDITIONS: Hand-Foot Syndrome; Breast Cancer
MeSH Terms: conditions — Hand-Foot Syndrome; Breast Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ice Plant Intensive Cream plus Standard Care (Experimental): This group receives a 30-minute nursing consultation on the standard treatment and on the use of the Ice Plant Intensive Cream for the prevention of hand-foot syndrome.
  Interventions: Other: Ice Plant Intensive Cream plus Standard Care
- Standard Care (Active Comparator): This group receives a 30-minute nursing consultation on the standard treatment for the prevention of hand-foot syndrome.
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Ice Plant Intensive Cream plus Standard Care — This group receives a 30-minute nursing consultation on the standard treatment according to the guideline "Supportive Therapy" for hand-foot syndrome and on the use of the Ice Plant Intensive Cream for the prevention of hand-foot syndrome. The nursing consultation on the standard treatment includes recommended basic measures for the prophylaxis of hand-foot syndrome such as the avoidance of mechanical stress and chemical irritants. In addition, treatment of pre-existing skin conditions is recommended. Furthermore, prophylaxis with urea-containing cream (5-10%) should be applied several times a day.
  Arms: Ice Plant Intensive Cream plus Standard Care
Other: Standard Care — This group receives a 30-minute nursing consultation on the standard treatment according to the guideline "Supportive Therapy" for hand-foot syndrome. The nursing consultation includes recommended basic measures for the prophylaxis of hand-foot syndrome such as the avoidance of mechanical stress and chemical irritants. In addition, treatment of pre-existing skin conditions is recommended. Furthermore, prophylaxis with urea-containing cream (5-10%) should be applied several times a day.
  Arms: Standard Care

SUMMARY:
The present pilot study investigates the feasibility of a prospective larger confirmatory study on the efficacy of Dr. Hauschka Med Ice Plant Intensive Cream for the prevention of hand-foot syndrome in patients with breast carcinoma undergoing therapy with doxorubicin and / or docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients
* Therapy with Doxorubicin and/or Docetaxel
* Karnofsky performance status scale > 80
* Informed consent

Exclusion Criteria:

* Patients with previous skin disease and/or polyneuropathy
* Intolerance or allergic reaction on at least one ingredient of Ice Plant Intensive Cream
* Already receiving chemotherapy
* Usage of Ice Plant Intensive Cream before trial
* Severe physical or psychological illness due to which the patient is not able to participate in the study
* Lack of German language skills

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Number of patients that can be recruited in a 9 months time period | 7 days after last chemotherapy cycle (each cycle is 3-4 weeks)
  The number of patients that can be recruited in a 9 months time period will be recorded in the study center
Proportion of potentially eligible patients that agree to participate in the study and thus to randomization | 7 days after last chemotherapy cycle (each cycle 3-4 weeks )
  The proportion of potentially eligible patients that agree to participate in the study and thus to randomization will be recorded in the study center
Proportion of randomized patients who leave the study early | 7 days after last chemotherapy cycle (each cycle is 3-4 weeks)
  The proportion of randomized patients who leave the study early will be recorded in the study center
Number of days in which the symptom diary was completed correctly | 7 days after last chemotherapy cycle (each cycle is 3-4 weeks)
  Symptoms will be collected daily in a symptom diary. The completeness of each patient diary will be assessed.
Number of days in which the intervention was carried out per protocol | 7 days after last chemotherapy cycle (each cycle is 3-4 weeks)
  The number of days in which the intervention was carried out and how often per day the intervention was carried out will be collected daily in a diary. The number of days in which the intervention was carried out will be assessed.

SECONDARY OUTCOMES:
Prevention of the hand-foot syndrome | From the start of chemotherapy to 7 days after the last chemotherapy cycle (daily diary) (each cycle is 3-4 weeks)
  Prevention of the hand-foot syndrome (WHO-scale daily rating)
Severity of the hand-foot syndrome | From the start of chemotherapy to 7 days after the last chemotherapy cycle (diary) (each cycle is 3-4 weeks)
  Severity of the hand-foot syndrome (WHO-scale daily rating)
Pain in hands and feet | From the start of chemotherapy to 7 days after the last chemotherapy cycle (diary) (each cycle is 3-4 weeks)
  Pain in hands and feet (Numerical Rating Scale daily rating)
Sensory disturbances in the hands and feet | From the start of chemotherapy to 7 days after the last chemotherapy cycle (diary) (each cycle is 3-4 weeks)
  Sensory disturbances in the hands and feet (Numerical Rating Scale daily rating)
Impairment of daily life due to the changes in the hands and feet | From the start of chemotherapy to 7 days after the last chemotherapy cycle (diary) (each cycle is 3-4 weeks)
  Impairment of daily life due to the changes in the hands and feet (Numerical Rating Scale daily rating)
Dermatology Life Quality Index (DLQI) questionnaire | 7 days after the first chemotherapy cycle (each cycle is 3-4 weeks)
  The DLQI provides information about changes over the course of therapy. It is a useful tool to determine the success of ongoing treatment. It is the most commonly used instrument in randomized controlled trials in dermatology.
Dermatology Life Quality Index (DLQI) questionnaire | 7 days after the third chemotherapy cycle (each cycle is 3-4 weeks)
  The DLQI provides information about changes over the course of therapy. It is a useful tool to determine the success of ongoing treatment. It is the most commonly used instrument in randomized controlled trials in dermatology.
Dermatology Life Quality Index (DLQI) questionnaire | 7 days after the last chemotherapy cycle "through study completion, an average of 1 year".(each cycle is 3-4 weeks)
  The DLQI provides information about changes over the course of therapy. It is a useful tool to determine the success of ongoing treatment. It is the most commonly used instrument in randomized controlled trials in dermatology.

CONTACTS AND LOCATIONS:
Locations (1):
- Robert-Bosch-Hospital, Stuttgart, Germany